CLINICAL TRIAL: NCT03128619
Title: A Phase Ib Trial Evaluating the Safety of Copanlisib, Letrozole, and Palbociclib in Metastatic Breast Cancer and Phase II Trial Comparing the Molecular Effects of Neoadjuvant Copanlisib in Combination With Palbociclib and Letrozole, vs. Copanlisib With Letrozole, vs. Palbociclib With Letrozole for Patients With Hormone Receptor Positive, HER2 Normal Breast Cancer
Brief Title: Copanlisib, Letrozole, and Palbociclib in Treating Patients With Hormone Receptor Positive HER2 Negative Stage I-IV Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Bayer (Industry); Translational Research in Oncology-U.S. Inc. (TRIO-US) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-001271; NCI-2017-00435 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-04-04; First posted 2017-04-25 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2021-04

CONDITIONS: Estrogen Receptor Positive; HER2/Neu Negative; Invasive Breast Carcinoma; Multifocal Breast Carcinoma; Postmenopausal; Progesterone Receptor Positive; Stage I Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — copanlisib; Letrozole; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (copanlisib, letrozole) (Experimental): PHASE II: Patients receive copanlisib (MTD) IV over 1 hour on days 1, 8, and 15 and letrozole PO continuously on days 1-28. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression, or unacceptable toxicity.
  Interventions: Drug: Copanlisib; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Other: Pharmacological Study
- Arm B (copanlisib, palbociclib, letrozole) (Experimental): PHASE II: Patients receive copanlisib (MTD) IV over 1 hour on days 1, 8, and 15, palbociclib PO QD on days 1-21, and letrozole PO continuously on days 1-28. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy of Breast; Drug: Copanlisib; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Drug: Palbociclib; Other: Pharmacological Study
- Arm C (copanlisib, palbociclib, letrozole) (Experimental): PHASE II: Patients receive palbociclib PO QD for days 1-14 of course 1 and letrozole PO continuously on days 1-14. Patients then undergo biopsy. Patients then receive copanlisib IV over 1 hour on days 1, 8, and 15 and letrozole PO continuously on days 1-28. Treatment with copanlisib (MTD) and letrozole repeats every 28 days for up to 3.5 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy of Breast; Drug: Copanlisib; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Drug: Palbociclib; Other: Pharmacological Study
- Phase Ib (copanlisib, palbociclib, letrozole) (Experimental): PHASE Ib: Patients with metastatic breast cancer receive copanlisib IV over 1 hour on days 1, 8, and 15, palbociclib PO QD on days 1-21, and letrozole PO continuously on days 1-28. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Copanlisib; Other: Laboratory Biomarker Analysis; Drug: Letrozole; Drug: Palbociclib; Other: Pharmacological Study

INTERVENTIONS:
Procedure: Biopsy of Breast — Undergo biopsy
  Other Names: Breast Biopsy
  Arms: Arm B (copanlisib, palbociclib, letrozole); Arm C (copanlisib, palbociclib, letrozole)
Drug: Copanlisib — Given IV
  Other Names: BAY 80-6946; PI3K Inhibitor BAY 80-6946
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
Drug: Palbociclib — Given PO
  Other Names: Ibrance; PD-0332991; PD-332991
  Arms: Arm B (copanlisib, palbociclib, letrozole); Arm C (copanlisib, palbociclib, letrozole); Phase Ib (copanlisib, palbociclib, letrozole)
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies side effects and best dose of copanlisib when given together with letrozole and palbociclib and to see how well they work in treating hormone receptor positive HER2 negative stage I-IV breast cancer. Copanlisib and palbociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs, such as letrozole, may lessen the amount of estrogen made by the body. Giving copanlisib, letrozole, and palbociclib may work better in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety, tolerability and to estimate the maximum tolerated dose (MTD) in a metastatic setting of the following combination: copanlisib + palbociclib + letrozole. (Phase Ib) II. Compare the biological activity of letrozole in combination with palbociclib, letrozole in combination with palbociclib and copanlisib, and letrozole in combination with copanlisib by assessing the percentage change from the baseline value in Ki67 expression after 2 weeks of therapy in non-metastatic breast cancer. (Phase II)

SECONDARY OBJECTIVES:

I. Evaluate the pathologic complete response (pCR) defined as absence of invasive cancer in the breast and sampled regional lymph nodes.

II. Evaluate the clinical objective response Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1.

III. Assess safety and tolerability. IV. Evaluate the pharmacokinetics of copanlisib when given in combination with letrozole, and palbociclib.

V. Measure the gene expression and/or biomarker changes that may be correlated with or predict biological, clinical, and pathologic response.

OUTLINE: This is a dose-escalation study of copanlisib.

PHASE Ib: Patients with metastatic breast cancer receive copanlisib intravenously (IV) over 1 hour on days 1, 8, and 15, palbociclib orally (PO) once daily (QD) on days 1-21, and letrozole PO continuously on days 1-28. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

PHASE II: After determination of MTD, subsequent non-metastatic breast cancer patients are randomized to 1 of 3 arms:

ARM A: Patients receive copanlisib (MTD) IV over 1 hour on days 1, 8, and 15 and letrozole PO continuously on days 1-28. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression, or unacceptable toxicity.

ARM B: Patients receive copanlisib (MTD) IV over 1 hour on days 1, 8, and 15, palbociclib PO QD on days 1-21, and letrozole PO continuously on days 1-28. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive palbociclib PO QD for days 1-14 of course 1 and letrozole PO continuously on days 1-14. Patients then undergo biopsy. Patients then receive copanlisib (MTD) IV over 1 hour on days 1, 8, and 15 and letrozole PO continuously on days 1-28. Treatment with copanlisib and letrozole repeats every 28 days for up to 3.5 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal (if female) defined as: 1) prior bilateral oophorectomy, 2) age 60 or over, or 3) < 60 years and amenorrheic for at least 12 months with follicle-stimulating hormone (FSH) and estradiol in the postmenopausal range per institutional parameters); use of luteinizing hormone-releasing hormone (LHRH) agonists to induce chemical ovarian ablation will not be allowed for this study
* Tumor is hormone receptor (HR)+ (estrogen receptor and/or progesterone receptor positive with at least 10% expression of either receptor by local immunohistochemical staining) and HER2 negative based on local assessment
* FOR PHASE Ib PORTION OF THE STUDY:
* Locally advanced/non-operable or metastatic breast cancer that has not been previously treated in the metastatic setting with systemic therapy (i.e. first line treatment)
* Measurable disease per RECIST 1.1
* FOR PHASE II PORTION OF THE STUDY:
* Clinical stage I (breast tumor >= 1.0 cm in diameter), stage II or stage III breast cancer (according to the American Joint Committee on Cancer [AJCC] Staging Manual, 7th Edition, 2010); multifocal disease is allowed if confined to 1 breast, as long as one tumor is at least 1 cm and meets all of the other inclusion criteria
* Breast cancer suitable for mandatory baseline core biopsy
* No prior systemic therapy or radiotherapy for currently-diagnosed invasive or noninvasive breast cancer
* FOR ALL PHASES (Ib AND II):
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets > 100 x 10^9/L
* Hemoglobin >= 8 g/dL (phase Ib) or >= 10 g/dL (for phase II portion)

  * For phase Ib portion only: patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator; however, initial study drug treatment must not begin earlier than the day of the erythrocyte transfusion
* Bilirubin =< 1.5 times the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 times ULN
* Subjects with Gilbert's syndrome, confirmed by genotyping or Invader UGTIA1 molecular assay prior to study entry, must have total bilirubin < 3.0 times ULN
* Serum creatinine =< 1.5 times ULN
* Lipase =< 1.5 x ULN
* International normalized ratio (INR) and partial thromboplastin time (PTT) < 1.5 x ULN
* Left ventricular ejection fraction (LVEF) >= 50%
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* FOR PHASE Ib ONLY:
* Early stage (curable) breast cancer
* FOR PHASE II ONLY:
* Metastatic breast cancer (local spread to axillary or internal mammary lymph nodes is permitted)
* Prior systemic therapy for invasive or non-invasive (DCIS) breast cancer
* Prior radiotherapy to the ipsilateral chest wall or breast for any malignancy
* Bilateral invasive breast cancer
* FOR ALL PHASES (Ib AND II): Inflammatory breast cancer
* FOR ALL PHASES (Ib AND II): Concurrent therapy with any other non-protocol anti-cancer therapy
* FOR ALL PHASES (Ib AND II): History of any other malignancy within the past 5 years, with the exception of non-melanoma skin cancer or carcinoma-in-situ of the cervix
* FOR ALL PHASES (Ib AND II): Concurrent diagnosis of pheochromocytoma
* FOR ALL PHASES (Ib AND II): Current therapy with raloxifene, tamoxifen, aromatase inhibitor, or other selective estrogen receptor modulator (SERM), either for osteoporosis or prevention of breast cancer; subjects must have discontinued therapies for at least 28 days prior to first baseline biopsy
* FOR ALL PHASES (Ib AND II): Concurrent treatment with postmenopausal hormone replacement therapy; prior treatment must be stopped for at least 28 days prior to first baseline biopsy
* FOR ALL PHASES (Ib AND II): Type I diabetes or patients on insulin therapy are not allowed; uncontrolled type II diabetes not allowed (glycosylated hemoglobin [HbA1c] > 7.5)
* FOR ALL PHASES (Ib AND II): Proteinuria of >= Common Terminology Criteria for Adverse Events (CTCAE) grade 3 as estimated by urine protein : creatinine ratio > 3.5 on a random urine sample
* FOR ALL PHASES (Ib AND II): Uncontrolled arterial hypertension despite optimal medical management
* FOR ALL PHASES (Ib AND II): Hepatitis B (HBV) or hepatitis C (HCV); all patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus laboratorial panel
* FOR ALL PHASES (Ib AND II): Known history of human immunodeficiency virus (HIV) infection
* FOR ALL PHASES (Ib AND II): Uncontrolled infection; active, clinically serious infections (> CTCAE grade 2)
* FOR ALL PHASES (Ib AND II): History of significant cardiac disease:

  * Congestive heart failure > New York Heart Association (NYHA) class 2
  * Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
  * Myocardial infarction less than 6 months before start of test drug
  * Anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* FOR ALL PHASES (Ib AND II): Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication
* FOR ALL PHASES (Ib AND II): Participants receiving anticoagulation therapy are not allowed
* FOR ALL PHASES (Ib AND II): Patients with evidence or history of bleeding diathesis; any hemorrhage or bleeding event >= CTCAE grade 3 within 4 weeks of start of study medication
* FOR ALL PHASES (Ib AND II): Blood or platelet transfusion within 7 days prior to treatment start
* FOR ALL PHASES (Ib AND II): Non-healing wound or ulcer
* FOR ALL PHASES (Ib AND II): History of, or current autoimmune disease
* FOR ALL PHASES (Ib AND II): Major surgical procedure or significant traumatic injury (as judged by the investigator) within 28 days before start of study medication, open biopsy within 7 days before start of study medication
* FOR ALL PHASES (Ib AND II): Patients with seizure disorder requiring medication
* FOR ALL PHASES (Ib AND II): Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
* FOR ALL PHASES (Ib AND II): Systemic continuous corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not allowed; patients may be using topical or inhaled corticosteroids; previous corticosteroid therapy must be stopped or reduced to the allowed dose at least 7 days prior to the first study drug administration; if a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose after the patient has signed the consent document
* FOR ALL PHASES (Ib AND II): History of having received an allogeneic bone marrow or organ transplant
* FOR ALL PHASES (Ib AND II): Chronic oxygen therapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Ki-67 expression defined as the percent of cells staining positive by validated central assay (Phase II) | Baseline to 2 weeks
  Will be evaluated on the log Ki-67 ratio scale. Primary analysis of this variable will utilize a linear model with treatment, PR status as fixed effects. The comparison of treatment arms will be based on the least squares mean (LSM) estimates and standard errors derived from this model. For descriptive purposes, LSM estimates and associated confidence intervals (CIs) will be back transformed to the geometric mean percent change scale. A second post-baseline evaluation of Ki67 expression will be performed following the completion of 4 months of treatment. Analysis of change from baseline to com
Incidence of dose-limiting toxicities (DLT) evaluated according to National Cancer Institute (NCI) CTCAE version 4.0 to determine MTD (Phase Ib) | Up to 112 days
  If >= 2 of 6 participants treated at a dose level experience DLTs, then the MTD will have been exceeded. Up to 3 additional patients may be entered at the lower dose level to obtain additional safety information (if only 3 participants were treated previously at that dose) to demonstrate that =< 1 of 6 patients experience DLT.

SECONDARY OUTCOMES:
Clinical objective response rate (ORR) evaluated by RECIST 1.1 using caliper measurements | Up to 1 month after surgery
  A responder is defined as any participant who exhibits a complete response (CR) or partial response (PR). The clinical response rate is estimated as the total number of CRs and PRs divided by the total number of participants randomized. Clinical ORR will be estimated and 95% exact CIs will be provided.
Gene expression and/or biomarker changes | Up to 1 month after surgery
  To compare the percent change in Ki67 expression from baseline to 2 weeks in the Ki67-evaluable population (expansion phase only).The Ki67 Evaluable Population will include all patients with a valid baseline Ki67 measurement of at least 5% and a valid 2-week measurement of any magnitude. This population will be used for the analysis of all Ki67-derived endpoints. All ki67 evaluable population will be correlated with pCR and clinical objective response.
Incidence of adverse events (AEs) evaluated according to NCI CTCAE version 4.0 | Up to 1 month after surgery
  Overall exposure to study drug, the numbers of patients completing each cycle and the dose intensity will be summarized using descriptive statistics. The number of patients with any dose adjustment will be presented for entire treatment period as well as for each cycle. The number of patients with dose reductions, dose delays, or dose omissions will also be summarized, as will the reasons for dose adjustments. AEs and severe AEs will be reported using a CTCAE version 4.0 terminology and severity.
pCR rate defined as the percentage of randomized patients with a pCR | Up to 1 month after surgery
  pCR is defined as the absence of invasive cancer in the breast and sampled regional lymph nodes. Pathology reports from definitive breast surgery will be collected.
The pharmacokinetic (PK) parameter - area under the plasma concentration-time curve (AUC) will be determined for copanlisib in arms A, B, and escalation dose levels. | At pre-infusion, 10 minutes, 1, 2, 3, and 5 hours after start of infusion on days 1 and 8, course 1 (Ib); at pre-infusion and 1 hour after start of infusion on day 1, course 1 and pre-infusion, 5-15 minutes, 1, and 1-1.5 hours on day 8, course 2 (II)
  PK sampling will be performed in all the participants to characterize the PK profile for copanlisib, its metabolite M-1 (and other metabolites) in combination with letrozole and palbociclib.
The pharmacokinetic (PK) parameter - Elimination half-life (t½) will be determined for copanlisib in arms A, B, and escalation dose levels. | At pre-infusion, 10 minutes, 1, 2, 3, and 5 hours after start of infusion on days 1 and 8, course 1 (Ib); at pre-infusion and 1 hour after start of infusion on day 1, course 1 and pre-infusion, 5-15 minutes, 1, and 1-1.5 hours on day 8, course 2 (II)
  PK sampling will be performed in all the participants to characterize the PK profile for copanlisib, its metabolite M-1 (and other metabolites) in combination with letrozole and palbociclib.
The pharmacokinetic (PK) parameter - Maximum plasma concentration (Cmax) will be determined for copanlisib in arms A, B, and escalation dose levels. | At pre-infusion, 10 minutes, 1, 2, 3, and 5 hours after start of infusion on days 1 and 8, course 1 (Ib); at pre-infusion and 1 hour after start of infusion on day 1, course 1 and pre-infusion, 5-15 minutes, 1, and 1-1.5 hours on day 8, course 2 (II)
  PK sampling will be performed in all the participants to characterize the PK profile for copanlisib, its metabolite M-1 (and other metabolites) in combination with letrozole and palbociclib.
The pharmacokinetic (PK) parameter - Minimum plasma concentration of BAY 80-694 will be determined for copanlisib in arms A, B, and escalation dose levels. | At pre-infusion, 10 minutes, 1, 2, 3, and 5 hours after start of infusion on days 1 and 8, course 1 (Ib); at pre-infusion and 1 hour after start of infusion on day 1, course 1 and pre-infusion, 5-15 minutes, 1, and 1-1.5 hours on day 8, course 2 (II)
  PK sampling will be performed in all the participants to characterize the PK profile for copanlisib, its metabolite M-1 (and other metabolites) in combination with letrozole and palbociclib.
The pharmacokinetic (PK) parameter - Time when Cmax occurs (Tmax) will be determined for copanlisib in arms A, B, and escalation dose levels. | At pre-infusion, 10 minutes, 1, 2, 3, and 5 hours after start of infusion on days 1 and 8, course 1 (Ib); at pre-infusion and 1 hour after start of infusion on day 1, course 1 and pre-infusion, 5-15 minutes, 1, and 1-1.5 hours on day 8, course 2 (II)
  PK sampling will be performed in all the participants to characterize the PK profile for copanlisib, its metabolite M-1 (and other metabolites) in combination with letrozole and palbociclib.
The pharmacokinetic (PK) parameter - Average plasma concentration at steady state (Cavg) will be determined for copanlisib in arms A, B, and escalation dose levels. | At pre-infusion, 10 minutes, 1, 2, 3, and 5 hours after start of infusion on days 1 and 8, course 1 (Ib); at pre-infusion and 1 hour after start of infusion on day 1, course 1 and pre-infusion, 5-15 minutes, 1, and 1-1.5 hours on day 8, course 2 (II)
  PK sampling will be performed in all the participants to characterize the PK profile for copanlisib, its metabolite M-1 (and other metabolites) in combination with letrozole and palbociclib.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hurvitz, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States